CLINICAL TRIAL: NCT06393504
Title: Healthcare Claims Database Study to Provide Safety Information on Maternal, Fetal and Infant Outcomes Among Women Exposed to QUVIVIQ (Daridorexant) During Pregnancy
Brief Title: Database Study to Provide Information on Pregnancy and Infant Outcomes Among Women Exposed to QUVIVIQ (Daridorexant)
Status: Active, not recruiting | Type: Observational
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Collaborators: Carelon Research (Other)
Responsible Party: Sponsor
Other Study IDs: ID-078A404
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Disorder
Keywords: Pregnancy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- QUVIVIQ-exposed group: Pregnant women with insomnia exposed to QUVIVIQ during pregnancy or within 5 half-lives prior to date of conception.
  Interventions: Drug: Daridorexant
- Active comparator group: Pregnant women with insomnia exposed to non-orexin receptor antagonist insomnia medications during pregnancy or within 5 half-lives of the respective insomnia medication prior to date of conception.
  Interventions: Drug: Non-orexin receptor antagonist insomnia medication
- Unexposed comparator group: Pregnant women with insomnia unexposed to insomnia medications during pregnancy and within 5 half-lives of any insomnia medication taken prior to date of conception.
  Interventions: Other: No insomnia medication

INTERVENTIONS:
Drug: Daridorexant — Daridorexant received during or shortly prior to pregnancy.
  Other Names: QUVIVIQ
  Groups: QUVIVIQ-exposed group
Drug: Non-orexin receptor antagonist insomnia medication — Non-orexin receptor antagonist insomnia medication received during or shortly prior to pregnancy.
  Groups: Active comparator group
Other: No insomnia medication — No insomnia medication received during or shortly prior to pregnancy.
  Groups: Unexposed comparator group

SUMMARY:
Healthcare claims database study to provide safety information on maternal, fetal and infant outcomes among women exposed to QUVIVIQ (daridorexant) during pregnancy

DETAILED DESCRIPTION:
This is a longitudinal observational cohort study using an electronic database of healthcare claims data. Safety information will be retrospectively collected from the database and pre-specified diagnostic codes will be used to identify pregnancy and infant outcomes. The study will include two phases, a patient accrual phase (Phase 1) and an analysis phase (Phase 2).

Descriptive statistics will be conducted to characterize the patient population and to support the interpretation of comparative analyses. Comparative analyses will be performed to estimate the effect of QUVIVIQ exposure during pregnancy on the study outcomes. Approximately 419 mother-infant pairs with exposure to QUVIVIQ and 1676 mother-infant pairs with exposure to non-orexin receptor antagonist insomnia medication are expected with a 1:4 ratio of exposed:active comparator patients.

Analysis of the prevalence of each specific pregnancy or infant outcome will comprise: (1) a comparison between women with insomnia exposed to QUVIVIQ during or shortly prior to pregnancy (QUVIVIQ-exposed group) and women with insomnia exposed to any non-orexin receptor antagonist insomnia medication during or shortly prior to pregnancy (active comparator group); (2) a comparison between women with insomnia exposed to QUVIVIQ during or shortly prior to pregnancy (QUVIVIQ-exposed group) and women with insomnia unexposed to any insomnia medication during or shortly prior to pregnancy (unexposed comparator group).

ELIGIBILITY:
1. Evidence of a singleton end of pregnancy event during the intake period.
2. ≥ 1 insomnia diagnosis during the period which begins 12 months prior to the date of conception and ends at the end of pregnancy.
3. Continuous medical and pharmacy insurance coverage during the period which begins 6 months prior to the date of conception and ends at the date of conception plus 40 weeks (equivalent to 42 gestational weeks).
4. Age 15 to 50 years at the date of conception.
5. No dispensing of known or suspected teratogenic medications during the period which begins 5 half lives of that medication prior to the date of conception and ends at the end of pregnancy.
6. No exposure to other orexin receptor antagonists during the exposure period, i.e., suvorexant, lemborexant, and any orexin receptor antagonists newly approved during the intake period.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women with an end of pregnancy event between 1 May 2022 and 31 May 2027 (called the "intake period") and a diagnosis of insomnia disorder are included in the base cohort, from which the exposure- and outcome-specific analytic cohorts will be created.
Sampling Method: Non-Probability Sample
Enrollment: 2095 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of major congenital malformations (MCMs) | From May 2022 to April 2028 (6 years)
  MCMs will be identified as pre-specified diagnostic codes for malformations included in the National Birth Defects Prevention Network's birth defects descriptions (identified through maternal and infant claims).
  MCMs with etiologies presumed not to be associated with drug exposure, such as chromosomal abnormalities, genetic syndromes, prematurity-related defects, and positional effects, will be excluded from the definition of MCMs.

SECONDARY OUTCOMES:
Prevalence of spontaneous abortions (SABs) | From May 2022 to April 2028 (6 years)
  An SAB is defined as the loss of an embryo before 20 gestational weeks (identified through maternal claims).
Prevalence of stillbirths (SBs) | From May 2022 to April 2028 (6 years)
  An SB is defined as the loss of a fetus at or after 20 gestational weeks (identified through maternal claims).
Prevalence of small for gestational age infants (SGAs) | From May 2022 to April 2028 (6 years)
  SGA is defined as birth weight less than or equal to the tenth percentile for gestational age (identified through maternal and infant claims).
Prevalence of preterm births (PTBs) | From May 2022 to April 2028 (6 years)
  PTB is defined as a live birth before 37 gestational weeks (identified through maternal and infant claims).
Prevalence of induced abortions (IABs) | From May 2022 to April 2028 (6 years)
  An IAB is defined as the elective termination of the pregnancy (identified through maternal claims).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Study Director, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Carelon Research, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No